CLINICAL TRIAL: NCT00313872
Title: Phase III Randomized Trial of Taxotere/Cisplatin Followed by FOLFIRI or the Reverse Sequence in Unresectable Gastric Cancer
Brief Title: Phase III Trial of DP Followed by FOLFIRI or the Reverse Sequence in Unresectable Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMC IRB 2005-03-044
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Gastric Cancer; Metastases
Keywords: gastric cancer; chemotherapy; irinotecan; docetaxel
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis | interventions — IFL protocol

ARMS (2):
- FOLFIRI (Experimental)
  Interventions: Drug: FOLFIRI
- DP (Experimental): D1 Taxotere 75 mg/m2 + D5W 200 mL IV over 1 hr, D1 Cisplatin 75 mg/m2 + NS 150mL MIV over 1hr
  D1 Irinotecan 150 mg/m2 + D5W 500mL MIV over 90 min D1 Leucovorin 100 mg/m2 + D5W 500mL MIV over 2hrs D1-2 5-FU 1500 mg/m2 + D5W 1000 ml CIV over 24 hrs (total 2doses) D1 atropine 0.3mg SQ before irinotecan
  Interventions: Drug: DP

INTERVENTIONS:
Drug: DP — D1 Taxotere 75 mg/m2 + D5W 200 mL IV over 1 hr D1 Cisplatin 75 mg/m2 + NS 150mL MIV over 1hr Pre & Post medication Dexamethasone 8mg PO D0 Night (X1) D1 immediately upon waking in the morning, 1 hour before infusion Taxotere, Night (X3) D0 NS 1500 mL IV overnight hydration D1 DNK2 1000 mL IV over 2 hours, pre & post hydration (if Mg <WNL, mix MgSO4 1 amp) 20% Mannitol 70 mL IV full dripping, 30 mins before cisplatin D2-D3 Dexamethasone 8 mg PO bid, D4-D5 Dexamethasone 4 mg PO bid every 3 weeks
  Arms: DP
Drug: FOLFIRI — FOLFIRI regimen D1 Irinotecan 150 mg/m2 + D5W 500mL MIV over 90 min D1 Leucovorin 100 mg/m2 + D5W 500mL MIV over 2hrs D1-2 5-FU 1500 mg/m2 + D5W 1000 ml CIV over 24 hrs (total 2doses) D1 atropine 0.3mg SQ before irinotecan
  Arms: FOLFIRI

SUMMARY:
To assess the optimal sequence of the palliative chemotherapy regimen (DP --> FOLFIRI vs FOLFIRI --> DP) in metastatic gastric cancer patients.

DETAILED DESCRIPTION:
Gastric cancer is the second leading cause of cancer death worldwide and is the most common malignancy in Korea. Metastatic gastric cancer remains a therapeutic challenge for medical oncologists due to poor prognosis. A recent phase III trial comparing docetaxel-cisplatin-5-FU (DCF) to the reference arm of cisplatin-5-FU (CF) showed a significant superiority of DCF in terms of survival, time-to-progression, and response rate. However, because DCF regimen was associated with high incidence of toxicities, the regimen has not yet been widely accepted as the standard first-line chemotherapy for gastric cancer patients. Thus, the optimum front-line chemotherapy regimen should be extensively investigated in these patients to improve survival.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic adenocarcinoma of the stomach
2. Age ≥ 18
3. Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
4. Life expectancy of at least 3 months
5. Adequate renal, liver, bone marrow functions
6. Adjuvant chemotherapy more than 12 months from the date of study entry
7. Written informed consent

Exclusion Criteria:

1. Active infection requiring antibiotics
2. Pregnant, lactating women
3. Brain metastasis
4. Systemic illness not appropriate for chemotherapy
5. Radiotherapy within 2 weeks before the study entry
6. Allergy to drugs used in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2003-05; Primary Completion 2009-06 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Second progress-free survival | 2years

SECONDARY OUTCOMES:
Toxicity, overall survival | 2years

CONTACTS AND LOCATIONS:
Overall Officials: Won Ki Kang, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea